CLINICAL TRIAL: NCT05961566
Title: Palate Volumetric Change Analysis Following Connective Tissue Graft Harvesting With and Without Donor Site Augmentation: Randomized Controlled Trial
Brief Title: Palatal Volumetric Change Analysis Following Connective Tissue Graft With and Without Donor Site Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hailey Bivens (Other)
Responsible Party: Sponsor-Investigator, Hailey Bivens, Co-Investigator, Texas A&M University
Organization: Texas A&M University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB2023-0028
Record Dates: First submitted 2023-07-16; First posted 2023-07-27 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-07

CONDITIONS: Recession, Gingival
Keywords: Subepithelial connective tissue graft; Collagen matrix; Collagen sponge; Soft tissue augmentation; Palatal volumetric change
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Individuals will be randomly assigned to be in the control group of the intervention group (Collagen matrix soft tissue augmentation).
Who Masked: Outcomes Assessor
Masking Description: Individuals computing the statistical analysis will be masked for which outcome was used. Surgeons and patients will only know which outcome will be used at time of surgery.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Individuals with no addition of intervention (collagen matrix) after harvesting from the palate for a subepithelial connective tissue graft.
- Collagen Matrix (Experimental): Individuals with the addition of the intervention (collagen matrix) after harvesting form the palate for a subepithelial connective tissue graft.
  Interventions: Device: Use of collagen matrix after subepithelial connective tissue graft harvest

INTERVENTIONS:
Device: Use of collagen matrix after subepithelial connective tissue graft harvest — A collagen matrix is placed under the overlying flap after the subepithelial connective tissue graft harvesting.
  Other Names: Helistat - collagen matrix group; Experimental
  Arms: Collagen Matrix

SUMMARY:
The goal of this randomized clinical trial is to compare whether soft tissue augmentation placed in the donor site following a gum graft harvesting leads to volumetric changes compared to non-augmented sites in the palate. The main questions it aims to answer are:

* Are there tissue thickness changes between the two groups (control group and augmentation group)?
* Are there volumetric changes in the donor site (palate) between the two groups in the short and long term? Participants will receive a gum graft and then based on what group they were randomly assigned, they will receive either a collagen matrix where the gum graft was taken (on the palate) or nothing will be placed.

Researchers will compare non-augmented sites with augmented sites to see if there is a change in tissue thickness and volume.

DETAILED DESCRIPTION:
The randomized controlled trial aims to investigate the potential effect of post-harvesting donor site augmentation on palatal volumetric changes following connective tissue graft harvesting.

The study investigation is a randomized controlled trial (RCT) that aims to have 20 participants in each group. The palatal thickness will be clinically assessed and a digital intraoral scan of the palate will be performed pre-operatively. A subepithelial connect tissue graft will then be harvested from the palate. Patients will then be randomly assigned to receive/not receive augmentation of the donor site, using a collagen sponge. Palatal thickness measurements and intraoral scans will be repeated at 2-, 4-, and 6-months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Demographic

  1. Age: 18-65 years old
  2. Gender: Any
  3. Race: Any
  4. Non-smoker: no use of any tobacco product or nicotine-replacement products in the last 5 years
* Medical History

  1. Physically and mentally healthy with no contraindications for periodontal surgery
  2. American Society of Anesthesiologists: ASA-I or ASA-II
* Dental history

  1. Periodontally healthy
  2. No history of surgical interventions in the palate
  3. No history of cleft lip/palate
  4. No history of orthodontic treatment involving the palate (palatal expansion).
* Other

  1. Patients requiring mucogingival surgery involving connective tissue graft harvesting from the palate.
  2. Patients who are able and willing to provide informed consent
  3. Patients who are able and willing to follow study appointments

Exclusion Criteria:

* i. Medical History

  1. Smokers or users of nicotine replacement products
  2. Patients with a contraindication, e.g., allergy, for any of the medications or materials used in the study (benzocaine, lidocaine, chlorhexidine rinse, ibuprofen, acetaminophen, Glycolon ® sutures, collagen sponge matrix)
  3. Patients with diabetes (glycemic level > 110mg/l and HbA1c > 6.5%)
  4. Drug or alcohol abuse history
  5. Pregnancy, lactation.
  6. Patients with a history of bisphosphonate therapy, radiotherapy in the head and neck region for malignancies, or chemotherapy for treatment of malignant tumors
  7. Coagulation disorders or other systemic conditions affecting surgical or wound healing process and gingival tissues, such as cancer, HIV, metabolic bone diseases etc.
  8. Medications affecting periodontal status in the previous 6 months
  9. Medications affecting surgical or wound healing process and gingival tissues, such as phenytoin, cyclosporine, dihydropyridines, etc.
* Dental

  1. Patients with any history of palatal surgery
  2. Patients with inadequate donor site anatomy
  3. Poor oral hygiene

     1. Full-mouth plaque ≥ 20%
     2. Bleeding scores > 10%
  4. Untreated periodontitis

     1. Pocket depths > 3mm with BOP
     2. No active periodontal disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Palatal Thickness Change | 2 months, 4 months, 6 months
  Initial palatal thickness of first and second surgery will be measured prior to each surgical incision with an endodontic reamer
Palatal Volume Change | 2 months, 4 months, 6 months
  Palatal volume change will be compared using an intraoral scan where the scans will be overlayed to compare differences is volume change.

CONTACTS AND LOCATIONS:
Overall Officials: Ying S Wang, DDS, MS, Principal Investigator — Texas A&M School of Dentistry
Locations (1):
- Texas A&M College of Dentistry, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No